CLINICAL TRIAL: NCT04989595
Title: Real-world Performance Study Testing an Algorithm to Predict the Future Bleeding Profile of Women After Insertion of Intrauterine Systems for Contraception
Brief Title: A Study to Learn More About How a Smartphone App Called MyIUS Predicts Future Menstrual Bleeding in Women After They Have Begun Using Intrauterine Birth Control Method (a Birth Control Device is Inserted Into a Woman's Uterus by Her Doctor)
Acronym: MyIUS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21424
Record Dates: First submitted 2021-07-20; First posted 2021-08-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Uterine Bleeding Profile Prediction
Keywords: Prevention of pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women_Kyleena
  Interventions: Device: MyIUS app
- Women_Jaydess
  Interventions: Device: MyIUS app
- Women_Mirena
  Interventions: Device: MyIUS app

INTERVENTIONS:
Device: MyIUS app — Data will be self-reported by participants through the MyIUS app.

SUMMARY:
Researchers are looking to learn more about future menstrual bleeding in women who have started using intrauterine contraception methods. "Intrauterine contraception" means that a device is inserted into a woman's uterus by her doctor. The device then releases a birth control treatment into the uterus.

Researchers have found that when women use intrauterine contraception, its effects on the menstrual cycle can cause changes to how often and for how long women will bleed. This is one of reasons women may stop using their intrauterine contraception.

So, the researchers in this study wanted to learn about a tool that can be used to predict future bleeding events. This tool was developed based on the results of previous clinical studies that researched menstrual bleeding. This tool is a smartphone application called MyIUS.

This study will include about 3,000 women who have recently had intrauterine contraception inserted and who use the MyIUS app.

There will be no visits with a study doctor in this study. After the intrauterine contraception has been inserted, the women will start to record any events of bleeding in the MyIUS app. After they have recorded events of bleeding for a total of 90 days, the MyIUS app will give a prediction of menstrual bleeding expected for the next 180 days. The women who sign the electronic informed consent form will continue to record their bleeding events for a total of 6 months.

The researchers will then collect this information. They will use this information to find out how well the MyIUS app can predict future menstrual bleeding.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate that the bleeding prediction algorithm which was developed and validated based on clinical trial data also works in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Insertion of Kyleena, Jaydess, or Mirena IUS
* Female (of legal age to provide electronic informed consent (eIC)) using the MyIUS app
* Submitted eIC to use all data documented in the MyIUS app

Exclusion Criteria:

- None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women (of legal age to provide electronic informed consent (eIC)) after insertion of Kyleena, Jaydess, or Mirena who use medical device software (MyIUS app) for bleeding profile prediction at day 90.
Sampling Method: Non-Probability Sample
Enrollment: 3045 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Accuracy of the bleeding intensity prediction algorithm in predicting one out of three intensity clusters | Up to 270 days
  Intensity clusters: bleeding, spotting, none

SECONDARY OUTCOMES:
Accuracy of the menstrual cycle regularity prediction algorithm | Up to 270 days
Difference in accuracy of the original prediction algorithm compared to the adapted algorithm on the collected real-world data | Up to 270 days

CONTACTS AND LOCATIONS:
Locations (6):
- Many Locations, Many Locations, Brazil
- Many Locations, Many Locations, Denmark
- Many Locations, Many Locations, Germany
- Many Locations, Many Locations, Mexico
- Many Locations, Many Locations, Spain
- Many Locations, Many Locations, Sweden

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.